CLINICAL TRIAL: NCT05600946
Title: Characterization of Dysmorphology in Subjects With Creatine Transporter Deficiency
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: McMaster University, Ontario, Canada (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001074; 001074-CH
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-05-02

CONDITIONS: Cognitive Disorder; Metabolic Disease; Autism Spectrum Disorder
Keywords: Developmental Delay; Autism Spectrum Disorder; Children; Natural History
MeSH Terms: conditions — Cognitive Dysfunction; Metabolic Diseases; Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Affected individuals that meet inclusion criteria

SUMMARY:
Background:

Creatine transporter deficiency (CTD) is a genetic disorder that mainly affects the brain in males. CTD causes intellectual disability that can be mild to severe. People with CTD may have seizures and behavioral issues. They may have slow growth and tire easily. CTD may sometimes be confused with autism or other disorders. Better diagnostics are needed. The study team in an NIH study noted that the faces of children with CTD can look similar. For this natural history study, an expert will examine photos of children with CTD. Any shared traits found might help to diagnose CTD.

Objective:

To look for shared facial features of children with CTD.

Eligibility: Males aged 2 to 40 years old with CTD who were in study 17-CH-0020.

Design:

Some participants in study 17-CH-0020 had pictures taken of their faces. The NIH study team wants to share these photos with a colleague in Canada. This person is an expert at evaluating how genetic disorders affect people s bodies.

Participant data collected during the study may also be sent to this expert. This data may include diagnostic images and results from lab tests.

Some children did not have their pictures taken during study 17-CH-0020. Parents are asked to take pictures of these children and send them to the study team. These photos can be sent to a secure portal. The photos can also be taken in-person during a clinic visit.

The photos may be printed in clinical study journals. But this is not required. Parents will be asked to sign a separate consent before the photos are published....

DETAILED DESCRIPTION:
Study Description:

The purpose of this study is to evaluate photographs of subjects enrolled in Creatine Natural History Study of Males with Creatine Transporter Deficiency (CTD) based on our observation that many of these subjects have common craniofacial features. This will involve the participation of an outside investigator who has significant expertise in dysmorphology. We seek to determine whether specific dysmorphic features exist in this population.

Objectives:

Primary Objective: To characterize the dysmorphic features in subjects with CTD

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patient is male and between 2-40 years of age, inclusive.
  2. Patient has genomic confirmation of a pathologic mutation in the SLC6A8 gene.
  3. Patient is able to complete study-related procedures within limitations imposed by condition under study.
  4. Patients parents/guardians/caregivers must provide written consent (informed consent) to study-related procedures, and if appropriate, the patient will provide an assent.

EXCLUSION CRITERIA:

1. Patient has had status epilepticus within 3 months of screening.
2. Patients has had a seizure that lasts 5 minutes or longer, and a second seizure without recovering consciousness from the first one, or if a person has repeated seizures for 30 minutes or longer.
3. Patient is unable to comply with the study procedures or has a clinical disease or laboratory abnormality that in the opinion of the investigator would potentially increase the risk of participation.

Ages: 2 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Creatine Transport Deficiency
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
dysmorphic features | 3 years
  To characterize the dysmorphic features in subjects with CTD

CONTACTS AND LOCATIONS:
Overall Officials: Laverne G Mensah, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001074-CH.html